CLINICAL TRIAL: NCT00971347
Title: Randomized Controlled Trial of Chewing Gum for Weight Loss
Brief Title: Chewing Gum for Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Wm. Wrigley Jr. Company (Industry)
Responsible Party: David B. Allison, PhD/Professor of Public Health, The University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 000354619
Record Dates: First submitted 2009-09-02; First posted 2009-09-03 (Estimated); Last update posted 2010-11-23 (Estimated); Status verified 2010-11

CONDITIONS: Obesity; Overweight; Weight Loss
Keywords: obesity; overweight; weight loss; randomized controlled trial; chewing gum
MeSH Terms: conditions — Obesity; Overweight; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nutrition brochure (Active Comparator): Control participants will receive only a nutrition brochure, Finding Your Way to a Healthier You, based on a USDHHS/USDA publication, Dietary Guidelines for Americans 2005.
  Interventions: Behavioral: nutrition brochure
- Chewing gum + nutrition brochure (Experimental): Participants in the experimental arm will be instructed to incorporate gum chewing in their diet with a goal of at least 90 minutes per day. The schedule is 20 minutes each after breakfast, lunch and dinner plus 10 minutes mid-morning, mid-afternoon and 1 to 2 hours after dinner. Experimental participants also will be told to chew gum instead of unplanned eating in response to hunger, cravings, preoccupation with eating, or negative feelings.
  Interventions: Other: Extra sugar-free chewing gum sticks; Behavioral: nutrition brochure

INTERVENTIONS:
Other: Extra sugar-free chewing gum sticks — 90 minutes chewing per day after meals; mid-morning and mid-afternoon; 1 to 2 hours after dinner; and in response to hunger, cravings, preoccupation with eating, or negative feelings in general throughout the day.
  Other Names: Extra sugar-free chewing gum
  Arms: Chewing gum + nutrition brochure
Behavioral: nutrition brochure — one-time at baseline visit
  Other Names: Finding Your Way to a Healthier You (GPO 001-000-04718-3)

SUMMARY:
This is a randomized controlled trial of the effects of chewing gum on body weight. The investigators will randomly assign 200 overweight or mildly obese adults to one of two groups. Participants must be otherwise healthy and ages 19-50. The control group will receive only printed information on optimal diet and increasing physical activity. The intervention group will be instructed to chew gum following meals and in place of snacks for a minimum of 90 minutes per day. The intervention group also will receive the same information on optimal diet and increasing physical activity as the control group. In this 8-week intervention, the primary outcome will be change in body weight, and secondary outcomes will be changes in body mass income (BMI), waist circumference, and blood pressure. The protocol includes 3 clinic visits to assess outcomes: baseline, 4 weeks after randomization, and 8 weeks after randomization. Adherence to the gum chewing protocol will be assessed at clinic visits and during 2 telephone calls at 2 weeks and 6 weeks post-randomization. The investigators' hypothesis is that gum-chewers will lose more weight than those who receive information only.

DETAILED DESCRIPTION:
In this randomized controlled trial of the effects of chewing gum on body weight, we will randomly assign 200 overweight or mildly obese, but otherwise healthy adults (men and women, ages 19 to 50), to one of two groups: 1) a control group, which will receive printed information on optimal diet and increasing physical activity only, or 2) an intervention group, in which participants will be instructed to chew gum following meals and in place of snacks for a minimum of 90 minutes per day, in addition to receiving the same information on optimal diet and increasing physical activity as the control group. In this 8-week intervention, the primary outcome will be change in body weight, and secondary outcomes will be changes in body mass income (BMI), waist circumference, and blood pressure. Outcome measures will be assessed in both groups via clinic visits at baseline, 4 weeks post-randomization, and 8 weeks post-randomization. Adherence to the gum chewing protocol will be assessed at the clinic visits, as well as during telephone contacts at 2 weeks and 6 weeks post-randomization. The effects of the chewing gum intervention will be assessed by analysis of covariance (ANCOVA), wherein treatment assignment is the independent variable; the outcome measures described above will serve as dependent variables; and pre-randomization factors such as age, sex, and baseline BMI will be used as covariates. Our hypothesis is that those randomized to the intervention group will lowe more weight than those randomized to the control group.

ELIGIBILITY:
Inclusion Criteria:

* 19 - 50 years of age
* BMI 25 - 35 kg/m2
* Non-diabetic; no previous history of diabetes
* Fasting glucose <126 mg/dL at recruitment
* Male or female
* Any race or ethnicity

Exclusion Criteria:

* Any major disease including:
* Active cancer or cancer requiring treatment < 2 years (except nonmelanoma skin cancer).
* Active or chronic infections including self-reported HIV and active tuberculosis.
* Active cardiovascular disease or event with hospitalization; or therapeutic procedures for treatment of heart disease <6 months; or New York Heart Association Functional Class >2 for congestive heart failure, stroke or transient ischemic attack < 6 months.
* Uncontrolled hypertension: ≥SBP 160 mm Hg or DBP ≥95 mm Hg on treatment.
* GI disease: self-reported chronic hepatitis or cirrhosis; alcoholic hepatitis or alcoholic pancreatitis < 12 months; inflammatory bowel disease treatment < 12 months; recent or significant abdominal surgery.
* Renal disease: serum creatinine ≥1.4 mg/dL (124 μmol/L) for men; ≥1.3 mg/dL (115 μmol/L) for women.
* Lung disease: chronic obstructive airway disease with use of oxygen.
* Diagnosed diabetes (type 1 or 2), fasting hyperglycemia (blood glucose ≥ 126 mg/dL), or use of any anti-diabetic medications.
* Uncompensated or uncontrolled psychiatric disease that would impede conduct of the trial or completion of procedures.
* Phenylketonuria.
* Temporomandibular joint disorders.
* < 16 natural, fully crowned, or restored teeth in a good state of repair.
* Inadequate oral hygiene.
* Sensitivity to flavors, sweeteners, or other ingredients in sugar-free chewing gum.
* Refusal to chew gum per study guidelines.
* Currently chewing ≥5 sticks of gum per week.
* Weight loss or gain of >10% in the past 6 months except post-partum weight loss.
* Current participation in any weight-reduction program.
* Current smoker or quit < 6 months.
* History of prior surgical procedure for weight control or liposuction.
* Unable or unwilling to give informed consent; unable to communicate with clinic staff; another household member is a participant or staff member in the trial; unwilling to accept randomization; current or anticipated participation in another intervention research project that would interfere with the intervention offered in the trial; likely to move away before trial completed; unable to walk 0.25 mile in 10 minutes.
* Currently pregnant or < 3 months post partum; currently nursing or within 6 weeks of having completed nursing; pregnancy anticipated during study; unwilling to report possible or confirmed pregnancies promptly during the trial; unwilling to take adequate contraceptive measures if potentially fertile.
* Brief Symptom Inventory score (Derogatis & Melisaratos, 1983) > 90th percentile.
* Any active use of illegal or illicit drugs or history of such use < 12 months. Excessive alcohol intake, acute or chronic: average consumption of 3+ alcohol containing beverages daily; consumption of 7+ alcoholic beverages within a 24-hr period <12 months; or other evidence available to clinic staff. Subject may still be considered eligible if, upon explanation, the clinic staff believe that the volunteer can and will limit future intake.
* This is a partial listing; complete list available from PIs.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2009-08; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
weight change in kg | 8 weeks

SECONDARY OUTCOMES:
Body mass index in kilograms per meter-squared | 8 weeks
waist circumference in cm | 8 weeks
blood pressure in mm of mercury | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David B. Allison, PhD, Principal Investigator — University of Alabama at Birmingham; James M. Shikany, DrPH, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham Division of Preventive Medicine, Birmingham, Alabama, United States